CLINICAL TRIAL: NCT00746681
Title: A Phase 2, 26 Week, Multicentre, Randomized Double Blind, Placebo-Controlled, Crossover Study Evaluating the Efficacy and Safety of Tolterodine, Pregabalin and a Tolterodine-Pregabalin Combination for Idiopathic Overactive Bladder
Brief Title: Investigation of Tolterodine, Pregabalin and a Tolterodine - Pregabalin Combination for the Treatment of Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A8881001
Record Dates: First submitted 2008-04-02; First posted 2008-09-04 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): Tolterodine SR 2 mg once daily combined with pregabalin 75 mg twice daily
  Interventions: Drug: Tolterodine & Pregabalin
- B (Active Comparator): Tolterodine SR 4 mg once daily
  Interventions: Drug: Tolterodine
- C (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- D (Experimental): Tolterodine SR 4 mg once daily combined with pregabalin 150 mg twice daily
  Interventions: Drug: Tolterodine & Pregabalin
- E (Experimental): Pregabalin 150 mg twice daily
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Tolterodine & Pregabalin — Tolterodine SR Oral, 2mg, once daily for 4 weeks Pregabalin, Oral, 75 mg, twice daily for 4 weeks
  Arms: A
Drug: Tolterodine — Tolterodine SR, Oral, 4 mg, once daily for 4 weeks
  Arms: B
Drug: Placebo — Placebo, Oral, twice daily for 4 weeks
  Arms: C
Drug: Tolterodine & Pregabalin — Tolterodine SR Oral, 4mg, once daily for 4 weeks Pregabalin, Oral, 150 mg, twice daily for 4 weeks
  Arms: D
Drug: Pregabalin — Pregabalin, Oral, 150 mg twice daily for 4 weeks
  Arms: E

SUMMARY:
Tolterodine is approved for use in the treatment of overactive bladder (OAB). The study is designed to a investigate whether pregabalin may have efficacy in OAB and whether the efficacy is altered when it is combined with tolterodine.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years Old
* Diagnosis of OAB (micturition frequency >/= 8 times per day; urinary urgency >/= 4 times per week)

Exclusion Criteria:

* Subjects with symptoms of overactive bladder for less than 6 months prior to randomization.
* Significant stress incontinence as determined by the investigator e.g. stress predominant mixed incontinence, positive cough provocation test.
* Subjects with any condition that would contraindicate the use of tolterodine or pregabalin, including: Uncontrolled narrow angle glaucoma; Urinary retention; Myasthenia gravis; Gastric retention; Severe ulcerative colitis; Toxic megacolon; Rare hereditary problems of galactose intolerance; Fructose intolerance; Sucrose-isomalate insufficiency; Lapp lactase deficiency; Glucose-galactose malabsorption.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2005-12; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change in mean voided volume per micturition (from baseline). | 4 weeks

SECONDARY OUTCOMES:
Percentage and absolute change in incontinence episode frequency after 4 weeks of treatment (for subjects with incontinence at baseline). | 4 Weeks
Percentage and absolute change in urgency episode frequency | 4 Weeks
Mean severity of urgency episodes | 4 Weeks
Percentage and absolute change in micturition frequency | 4 Weeks
Percentage and absolute change in normalized micturition frequency (NMF) | 4 Weeks
Patient perception of their urinary urgency (using the OAB-q symptom severity scale) | 4 Weeks
Patient perception of Health Related Quality of Life (using the OAB-q SF HRQL scale) | 4 Weeks
Patient Perception of Bladder Condition (PPBC) scale | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Czechia (4):
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha 4 - Krc
  - Pfizer Investigational Site, Ústí nad Labem
- Lithuania (2):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Vilnius
- Norway (3):
  - Pfizer Investigational Site, Haugesund
  - Pfizer Investigational Site, Moelv
  - Pfizer Investigational Site, Trondheim
- Slovakia (4):
  - Pfizer Investigational Site, Martin, Slovakia
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Skalica
- Sweden (3):
  - Pfizer Investigational Site, Luleå
  - Pfizer Investigational Site, Norrköping
  - Pfizer Investigational Site, Stockholm
- United Kingdom (4):
  - Pfizer Investigational Site, Dundee, Tayside
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Plymouth

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8881001&StudyName=Investigation%20of%20tolterodine%2C%20pregabalin%20and%20a%20tolterodine%20-%20pregabalin%20combination%20for%20the%20treatment%20of%20overactive%20bladder.